CLINICAL TRIAL: NCT02909712
Title: Cardiac Safety of Dihydroartemisinin-Piperaquine Amongst Pregnant Women in Tanzania
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Kilimanjaro Christian Medical Centre, Tanzania (Other); National Institute for Medical Research, Tanzania (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: ITDCZF16
Record Dates: First submitted 2016-09-05; First posted 2016-09-21 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2020-01

CONDITIONS: Malaria; Pregnancy Malaria; Cardiotoxicity; Cardiac Safety; Parasitemia
Keywords: Sub-Saharan Africa; Dihydroartemisinin; Piperaquine; Sulphadoxine-Pyrimethamine; Antimalarials
MeSH Terms: conditions — Malaria; Cardiotoxicity; Parasitemia | interventions — fanasil, pyrimethamine drug combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sulfadoxine-pyrimethamine (SP) (Active Comparator): * Group 1 (50 CareStart™ RDT-positive women)
  * Group 2 (50 CareStart™ RDT-negative women)
  These 100 women will have an ECG exam, provide blood for microscopy and molecular analysis, and receive SP on day 0. On days 7, 14, 21, and 28 women will provide blood for microscopy and molecular analysis.
  Interventions: Drug: sulfadoxine-pyrimethamine (SP)
- dihydroartemisinin-piperaquine (DHA-PQP) (Experimental): * Group 3 (50 CareStart™ RDT-positive women)
  * Group 4 (50 CareStart™ RDT-negative women)
  These 100 women will have an ECG exam, provide blood for microscopy, molecular, and PK analysis, and receive DHA-PQP day 0. On day 1, women will receive dose 2. On day 2, women will have an ECG exam, begin Holter monitoring, provide blood for PK analysis, and receive dose 3. Blood for PK analysis will be drawn at 4, 5, and 6 hours following dose 3. An ECG exam will be conducted during this period and, again, on day 7. On days 7, 14, 21, and 28, women will provide blood for microscopy and molecular analysis.
  Interventions: Drug: dihydroartemisinin-piperaquine (DHA-PQP)

INTERVENTIONS:
Drug: sulfadoxine-pyrimethamine (SP) — Women in Groups 1 and 2 will be provided the following SP regimen as directly observed therapy:
  3 tablets total of 500 mg sulphadoxine and 25 mg pyrimethamine; 1 day of dosing.
  Other Names: Fansidar / Akacia Healthcare Ltd (South Africa)
  Arms: sulfadoxine-pyrimethamine (SP)
Drug: dihydroartemisinin-piperaquine (DHA-PQP) — Women in Groups 3 and 4 will be provided the following DHA-PQP regimen as directly observed therapy 3 tablets of 40 mg dihydroartemisinin and 320 mg piperaquine daily; 9 tablets total; 3 days of dosing.
  Other Names: Eurartesim / Sigma-Tau (Italy)
  Arms: dihydroartemisinin-piperaquine (DHA-PQP)

SUMMARY:
Sulfadoxine-pyrimethamine (SP) is currently recommended by the World Health Organization for use as intermittent preventive treatment against malaria in pregnancy (IPTp) in areas of moderate to high malaria transmission. However, in some locales malaria parasites have lost sensitivity to SP, compromising its protective effect. Dihydroartemisinin-piperaquine (DP) is a candidate replacement for SP. This trial is designed to confirm the cardio-safety of DP compared to SP amongst pregnant women in Tanzania.

DETAILED DESCRIPTION:
The trial hypothesis is that DP will increase the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle, a phenomenon referred to as QT prolongation, in the study population. However, if QT prolongation is observed, it is expected to be time-limited and of no clinical consequence.

The QT interval, measured in milliseconds (MS) will be corrected (QTc) to account for natural heart rate (HR) extremes. The Fridericia formula will also be used to correct (QTcF) for variation in cardio-contraction. As part of the electrocardiogram (ECG), the period from the beginning of the P wave to the beginning of the QRS complex (PR interval) will be measured, as well as the ST-segment which connects the QRS complex and the T wave.

Prolongation of the QT interval will be estimated when peak drug-concentrations are most likely to be found in the peripheral blood as measured using pharmacokinetic (PK) techniques. Polymerase chain reaction (PCR) methods will be used for genetic sequencing of molecular markers (A581G) associated with malaria parasite drug resistance to SP. The rapid diagnostic test (RDT) CareStart™ will be used to screen pregnant women attending antenatal care.

ELIGIBILITY:
Inclusion Criteria:

1. Participant presents for antenatal care at the district hospital.
2. Participant is between 18 years and 34 years of age.
3. Participant currently lives within the pre-defined catchment area of the district hospital.
4. Participant will remain within the same area through to the post-partum visit.
5. Participant agrees to deliver her child at the district hospital.
6. Participant agrees to a post-partum visit at her residence or at the district hospital.
7. Participant has no apparent severe infection or any condition that requires hospitalization.
8. Participant is not currently enrolled in another study.
9. Participant is not known to have heart disease or a known cardiac ailment.
10. Participant reports having taken no medication in the previous 28 days.
11. Participant reports having no known allergy to the study drugs or any sulphonamides.
12. Participant agrees to remain under observation for 3 hours at the district hospital and to abstain from food ingestion during the observation period in keeping with the European Medicines Agency product information for dosing with dihydroartemisinin-piperaquine.
13. Participant is willing to undergo all study procedures including sonography, ECG testing, and to provide blood samples for malaria microscopy and pharmacokinetic analysis.
14. Participant agrees to human immunodeficiency virus (HIV) testing regardless of prior results and no matter how recent.
15. Participant is not severely anaemic (haemoglobin concentration > 5g/dL).
16. Participant provides written consent.
17. Participant has an axillary temperature < 37.5 Celsius.
18. Participant is pregnant with a singleton determined by sonography.
19. Participant is between 16 and 35 weeks gestation determined by sonography.

Exclusion Criteria:

1. Participant is younger than 18 years of age and older than 35 years of age.
2. Participant does not currently live within the pre-defined catchment area of district hospital.
3. Participant will not remain within the same area through to the post-partum visit.
4. Participant does not agree to deliver her child at the district hospital.
5. Participant does not agree to a post-partum visit at her residence or at the district hospital.
6. Participant has a severe infection or any condition that requires hospitalization.
7. Participant is currently enrolled in another study.
8. Participant is known to have heart disease or known cardiac ailment.
9. Participant reports having taken any medication in the previous 28 days.
10. Participant reports having an allergy to the study drugs or any sulphonamides.
11. Participant does not agree to abstain from food ingestion during the observation period after dosing.
12. Participant does not agree to remain under observation at the district hospital 3 hours after dosing has occurred.
13. Participant does not agree or is unwilling to undergo all study procedures including sonography, ECG testing, and to provide blood samples for malaria microscopy (and treatment group assignment) and pharmacokinetic analysis.
14. Participant does not agree to HIV testing or is diagnosed as HIV-positive during screening,
15. Participant is not severely anaemic (haemoglobin concentration > 5g/dL).
16. Participant does not provide written consent.
17. Participant has an axillary temperature > 37.5 Celsius or is symptomatic for malaria.
18. Participant is carrying a multiple pregnancy (e.g. twins).
19. Participant is between < 16 weeks and > 36 weeks gestation.
20. Participant has a QTc > 450 milliseconds.
21. Participant has a heart rate < 40 beats per minute.

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 201 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Mean QTcF/QTcB change from baseline and proportion of pregnant women treated with DHA-PQP who experienced changes in RR, HR, PR, QRS, QT, QTcF and QTcB measurements from Day 0 pre-dose to Day 2 post-dose. | Measured on day 2 post-dose
Mean QTcF/QTcB change from baseline and proportion of pregnant women treated with DHA-PQP who experience changes in QT, QTcF and QTcB measurements from Day 0 pre-dose to Day 7. | Measured on day 7 post-dose

SECONDARY OUTCOMES:
Proportion of pregnant women treated with DHA-PQP/SP with and without asymptomatic parasitaemia who experienced clinical symptoms that could be related with a cardiac arrhythmia. | Measured on day 28 post-dose
  Clinical assessment
Mean QTcF/QTcB change from baseline and proportion of pregnant women treated with SP who experience changes in QT, QTcF and QTcB measurements from Day 0 pre-dose to Day 7 | Measured on day 7 post-dose
  Electrocardiography
Comparative analysis of the QT changes from Day 0 pre-dose to Day 7 post first dosing in pregnant women given DHA-PQP versus SP | Measured on day 7 post-dose
  Electrocardiography
Analysis of values and changes from baseline for the other electrocardiogram (ECG) parameters (RR, HR, PR, QRS) in pregnant women given DHA-PQP or SP | Measured on day 7 post-dose
  Electrocardiography
Adequate Parasitological Responses (APR) at Days 7, 14, 21 and 28 post-dose, PCR-Corrected and uncorrected | Measured on day 28 post-dose
  Efficacy
Proportion of participants in Groups 1-4 with parasites at Days 0, 7, 14, 21 and 28 that carry the 581G and/or K540E mutations associated with SP resistance | Measured on days 28 post-dose
  Parasite resistance

CONTACTS AND LOCATIONS:
Overall Officials: R. Matthew Chico, MPH, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Jacklin Mosha, MBBS, MSc, PhD, Principal Investigator — Kilimanjaro Christian Medical College
Locations (1):
- Handeni District Hospital, Handeni, Tanga, Tanzania

IPD SHARING:
Plan to Share IPD: No
Results will be published in a peer-reviewed journal

REFERENCES:
- [Background] Food and Drug Administration, HHS. International Conference on Harmonisation; guidance on E14 Clinical Evaluation of QT/QTc Interval Prolongation and Proarrhythmic Potential for Non-Antiarrhythmic Drugs; availability. Notice. Fed Regist. 2005 Oct 20;70(202):61134-5. PMID 16237860